CLINICAL TRIAL: NCT05398133
Title: Phenotype Assessment of Blood and Airway Eosinophils in Patients With COPD and Asthma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Other Study IDs: MB/M/15(31)
Record Dates: First submitted 2022-05-19; First posted 2022-05-31 (Actual); Last update posted 2022-05-31 (Actual); Status verified 2022-05

CONDITIONS: COPD Asthma; Eosinophilic Asthma
Keywords: eosinophil; COPD; asthma
MeSH Terms: conditions — Pulmonary Eosinophilia; Pulmonary Disease, Chronic Obstructive; Asthma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COPD patients
- asthma patients
- control subjects

SUMMARY:
Around 1/3 of patients with COPD have elevated eosinophil levels. However, the role of eosinophils in COPD has not been yet understood and is probably different in COPD and in asthma. The aim of this study was to assess the expression of selected surface markers on eosinophils and to assess the gene expression in eosinophils in COPD and asthma patients. We are planning to enrol 12 COPD, 12 asthma and 12 control subjects. Patients will undergo routine clinical assessment, spirometry, blood sampling and sputum induction. Eosinophils will be isolated from blood and sputum. Surface markers on eosinophils will be assessed in flow cytometry, gene expression will be assessed by RNAseq.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of COPD according to GOLD 2019 or asthma according to GINA 2021
* Peripheral blood eosinophil count ≥ 100 / μL
* Age ≥40 years (COPD), ≥18 years (asthma)
* History of cigarette smoking: ≥10 pack-years (for COPD)
* Stable disease period (at least 3 months without exacerbation)
* Exclusion of parasitic diseases
* Informed consent to participate in the study

Exclusion Criteria:

* COPD and asthma overlap
* Use of systemic corticosteroids in the 3 months prior to the study
* Respiratory infection or exacerbation in the 3 months prior to the study
* Acute and chronic respiratory failure
* Concomitant diagnoses: systemic connective tissue diseases, malignant neoplasms, severe and / or uncontrolled cardiovascular diseases
* Use of immunosuppressive or immunomodulating drugs in the 3 months preceding the study
* Contraindications to sputum induction
* No consent to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: COPD and asthma patients fulfilling the inclusion and exclusion criteria will be recruited from the outpatient clinic.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-06 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
expression of surface markers | performed up to 3 months after blood and sputum collection
  expression of CD125, CD62L, CD66b, CD193, CD11b, CD14

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Warsaw, Banacha Hospital, Warsaw, Poland

IPD SHARING:
Plan to Share IPD: No